CLINICAL TRIAL: NCT04309565
Title: Transitions Clinic Network: Post Incarceration Addiction Treatment, Healthcare, and Social Support
Acronym: TCN-PATHS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of North Carolina (Other); University of Puerto Rico (Other); University of Rochester (Other); University of Miami (Other); University of California, San Francisco (Other); University of Connecticut (Other); Albert Einstein College of Medicine (Other); Hennepin Healthcare Research Institute (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2000027469; 1UG1DA050072-01 (NIH)
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Opioid Addiction
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Hybrid type I effectiveness-implementation trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Primary Care (Active Comparator): Those randomized to the standard primary care arm will be referred to primary care and community Opioid Treatment Program (OTP). Participants may receive buprenorphine or Extended-release naltrexone (XR-NTX) through primary care or with a community addiction treatment provider.
  Interventions: Behavioral: Standard Primary Care
- Transitions Clinic Network Primary Care (Experimental): Transitions Clinic Network (TCN)- participants in this arm will be referred to a TCN program for primary care and community Opioid Treatment Program (OTP). All TCN programs have the ability to prescribe buprenorphine and Extended-release naltrexone (XR-NTX) and assist with referrals to methadone. The primary features of the TCN include (1) primary care and onsite MOUD or referral to community treatment when indicated, (2) addressing social determinants of OUD and care coordination through a Community Health Worker (CHW), and (3) addressing the discrimination and stigma that exist based on incarceration.
  Interventions: Behavioral: Transitions Clinic Network Primary Care

INTERVENTIONS:
Behavioral: Transitions Clinic Network Primary Care — Transitions Clinic Network (TCN)- participants in this arm will be referred to a TCN program for primary care and community Opioid Treatment Program (OTP). All TCN programs have the ability to prescribe buprenorphine and Extended-release naltrexone (XR-NTX) and assist with referrals to methadone. The primary features of the TCN include (1) primary care and onsite MOUD or referral to community treatment when indicated, (2) addressing social determinants of OUD and care coordination through a Community Health Worker (CHW), and (3) addressing the discrimination and stigma that exist based on incarceration.
  Arms: Transitions Clinic Network Primary Care
Behavioral: Standard Primary Care — Those randomized to the standard primary care arm will be referred to primary care and community Opioid Treatment Program (OTP). Participants may receive buprenorphine or Extended-release naltrexone (XR-NTX) through primary care or with a community addiction treatment provider.
  Arms: Standard Primary Care

SUMMARY:
TCN PATHS will recruit an anticipated 400 participants who are prescribed MOUD who are released from detention facilities. Each individual will be randomized to either 1) standard primary care (SPC) or 2) a Transitions Clinic Network (TCN) program primary care. Participants will be followed for a year and complete surveys at baseline and at month 1, 3, 6, 9, and 12. At each of these points research staff will confirm MOUD status. Urine drug screenings will be completed at baseline, month 1, 6, and 12 if the participant is not incarcerated. When possible, research staff will collect electronic health records.

DETAILED DESCRIPTION:
Purpose: The overall objective of this study is to assess whether the Transitions Clinic Network (TCN) program, which provides enhanced primary care and opioid use disorder (OUD) treatment for people recently released from incarceration, improves measures in the opioid treatment cascade compared to referral to standard primary care.

Participants: An anticipated 400 individuals currently receiving medications for OUD released from eight local jails (Durham, NC; Minneapolis, MN; Bronx, NY; Bridgeport and Niantic, CT; and Bayamón and Ponce, Puerto Rico)

Procedures: This is a hybrid type I effectiveness-implementation trial will randomize an anticipated 400 participants to one of two treatment conditions: TCN or standard primary care. People will complete the enrollment process while in jail (recruitment, screening, consent, baseline assessments, and randomization). Due to COVID-19 restrictions some jails are limiting researcher assess to people and some of our sites may enroll participants once they are released, this is referred to as a community enrollment. Post participants will meet with research assistants for a structured interview and urine toxicology screening at 1, 6, and 12 months, and a phone interview at months 3 and 9. 120 people will be selected to participate in Intensive Longitudinal Assessment (ILA) to access both the acceptability and appropriateness of the TCN intervention and the multi-level facilitators and barriers of OUD treatment engagement in the first 30 days following release from incarceration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English and Spanish-speaking,
* Meeting current DSM-5 criteria for OUD

Exclusion Criteria:

* acutely psychotic, suicidal or homicidal,
* require prescription opioids for acute pain, chronic pain or palliative care without OUD,
* have a planned relocation that makes it unlikely they would be able to complete the study and follow-up assessments,
* have a primary care provider that they already have established care with in the community,
* women of child-bearing age will be excluded if they are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Engagement in opioid use disorder (OUD) treatment | 30 days following jail release
  The primary study outcome will be engagement in OUD treatment within 30 days of jail release, defined as treatment consistent with the American Society of Addiction Medicine's levels of care (1-4), which allows for a range of treatments and clinical settings consistent with patient's needs and preference (e.g., office-based providers of buprenorphine or naltrexone, OTPs, or intensive outpatient, inpatient, or residential treatments). Patients do not need to be receiving methadone, buprenorphine, or naltrexone formulations (MOUD) to be considered engaged in OUD treatment. This will be measured based on questions about engagement in OUD treatment. These responses will be used to calculate a count of participants engaged in OUD treatment. As appropriate, this information will be confirmed in the electronic health record or with the addiction treatment facilities after obtaining a signed release.
Retention in OUD treatment | 12 months following jail release
  Retention in community OUD treatment will defined in accordance with the American Society of Addiction Medicine's levels of care (1-4), which allows for a range of treatments and clinical settings consistent with patient's needs and preference (e.g., office-based providers of buprenorphine or naltrexone, OTPs, or intensive outpatient, inpatient, or residential treatments). Patients do not need to be receiving MOUD to be considered retained in OUD treatment. Consistent with our prior research, this will be measured based on a Yes/No question about engagement in OUD treatment from the Treatment Services Review (TSR). These responses will be used to calculate a count of participants engaged in OUD treatment. As appropriate, this information will be confirmed in the electronic health record or with the addiction treatment facilities after obtaining a signed release. Re-incarceration (and resumption of MOUD in jail) will not count as retained in community OUD treatment.
Retention on medication for OUD (MOUD) | 12 months following initial jail release
  Retention on MOUD will be defined as receipt of any of the 3 FDA approved medications for OUD (methadone, buprenorphine, naltrexone) within 7 days of the index date (release from jail/interview date) regardless of what MOUD participants were on at baseline prior to release. This measure will be collected by using self report and as appropriate, will confirm self-report in the electronic health record or with the addiction treatment facilities after obtaining a signed release.
Percent days of illicit opioid use | 12 months following initial jail release
  Investigators will measure percent days of illicit opioid use during study time frames. Investigators will measure this by asking the participant how many days during the study time frame have they used illicit opioids. A urine toxicology that is positive for illicit opioids on testing will count as three days of using illicit opioids. Using the data from the

SECONDARY OUTCOMES:
Retention in primary care | 12 months following jail release
  Retention in primary care which is defined as 2 or more visits to primary care in twelve months. Participants will be asked to self-report the number of visits and this data will be used to count the number of participants retained in primary care.
Overdose | 12 months following initial jail release
  Participants will be asked about overdose events using self-report, when applicable, be supplemented by data from the electronic health record which will indicate visits to the emergency department and hospitalizations for overdose. In at least four TCN program sites, investigators will have access to administrative payer data (Medicaid) where investigators will be able to examine time to overdose as a secondary outcome. This data will be used to calculate a count of participants experiencing an overdose event
Time to Overdose | 12 months following initial jail release
  In at least four of the six TCN program sites, investigators will have access to administrative payer data (Medicaid) where investigators will be able to examine time to overdose as a secondary outcome. This data will be used to calculate time to overdose for each participant for each overdose event.
Death | 12 months following initial jail release
  Participant death will be collected using the electronic health record. In at least four of the six TCN program sites, investigators will have access to vital statistics data where survival analyses will be conducting with mortality as a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Wang, MD, Principal Investigator — Yale University
Locations (5):
- United States (4):
  - Yale, New Haven, Connecticut
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Albert Einstein College of Medicine, The Bronx, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howell BA, Puglisi L, Clark K, Albizu-Garcia C, Ashkin E, Booth T, Brinkley-Rubinstein L, Fiellin DA, Fox AD, Maurer KF, Lin HJ, McCollister K, Murphy S, Morse DS, Shavit S, Wang K, Winkelman T, Wang EA. The Transitions Clinic Network: Post Incarceration Addiction Treatment, Healthcare, and Social Support (TCN-PATHS): A hybrid type-1 effectiveness trial of enhanced primary care to improve opioid use disorder treatment outcomes following release from jail. J Subst Abuse Treat. 2021 Sep;128:108315. doi: 10.1016/j.jsat.2021.108315. Epub 2021 Jan 29. PMID 33583610